CLINICAL TRIAL: NCT05893901
Title: Impact of Food-to-Food Fortified Cereal Products on Diet Quality in Rural Niger Villages
Acronym: NigerMPS
Status: Completed | Type: Observational
Sponsor: Purdue University (Other)
Responsible Party: Principal Investigator, Bruce R. Hamaker, Principal Investigator / Distinguished professor, Purdue University
Other Study IDs: IRB-2022-571
Record Dates: First submitted 2023-05-30; First posted 2023-06-08 (Actual); Last update posted 2023-07-11 (Actual); Status verified 2023-07

CONDITIONS: Vitamin A Deficiency; Iron-deficiency
MeSH Terms: conditions — Vitamin A Deficiency; Anemia, Iron-Deficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Consumers of cereal products: Caregivers with children under 5 years of age who are consumer of cereal products in the Maradi, Falwell and Tera areas in Niger.

SUMMARY:
The primary hypothesis is that introduction of food-to-food fortified products through a rural Hub-and-Spoke incubator system contributes to an improved food environment and availability of micronutrients to these communities. A secondary hypothesis is that the influence of the rural Spokes can serve to enhance rural food environments through creation of secondary rural spokes that disseminate improved food-to-food fortified products.

The overall hypothesis is that a product designed with optimized nutritional characteristics, based on consumer preferences and leveraging local nutrient dense ingredients, can successfully deliver nutrition through sustainable market-driven approaches.

DETAILED DESCRIPTION:
Study Summary: Over the years our group has developed a Hub-and-Spoke incubator system to facilitate technology transfer and enable production, marketing, and sales of nutritionally improved cereal products in rural Niger. These efforts have led to the introduction of products developed using food-to-food fortification technology (FtFF). Examples of this include addition of moringa, carrot, cowpea, baobab powders to flours made with indigenous whole grains such as millet or sorghum. This technology leverages local nutrient dense plants to fortify cereal product traditionally consumed as porridges. These products are closely aligned to Corn-Soy Blends that are provided by international aid groups and dispensed/distributed through health centers at the village level. While these products provide a more complete nutritional profile for growing children and their families, their acceptability by children not always good and sustainability is poor as they are donor supported. Efforts to enhance the local community's food security and enhance nutritional quality of diets through local production and sales of FtFF products is key to developing sustainable improvements in local diets and nutrient availability. The investigators believe that the presence of Hub and Spoke incubator is critical to the success of these efforts, but data is needed to confirm their impact on the local food environment.

Study procedures:

Participants will be approached/recruited by research assistants (enumerators) in local markets and at sales locations. Potential participants will be approached and consented if they agree to join the study at the time of recruitment. Research assistants will read the consent form to the participants and ensure they understand it.

During the consumer interview, the investigators will be collecting the following information:

Consumer socioeconomics (for all) - this includes sex and age of each family member (no names or birth dates), and education level of the respondent Modified Food Frequency Questionnaire (for all) Diet Diversity Questionnaire - focus on pearl millet consumption (for all) Product specific questionnaire (for purchasers only)

* Product use: time of day, people in the household
* Product attributes they found most attractive
* 5-point-like scale: appearance, aroma, texture, taste.
* Overall convenience of flour product
* If small children were fed product, did they like it?
* Did other children like it?
* What did it replace?

ELIGIBILITY:
Inclusion Criteria:

* Adults (>18 years of age), with child(ren) 5 years of age living in the household.

Exclusion Criteria:

* No children under 5 y of age living in the household.
* Not a caregiver for the children in the household.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This study collected data about dietary habits for children and the household they lived. Adult caregivers were approached and provided the relevant information.
Sampling Method: Probability Sample
Enrollment: 3600 (Actual)
Dates: Start 2023-03-13 (Actual); Primary Completion 2023-05-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Assessment of staple intake in urban Nigerien households and children | 3 months
  A quantitative, modified food frequency questionnaire (FFQ) will be used to assess consumption of starch rich staples (rice, wheat, corn sorghum, millet, fonio, potatoes, cassava, yams) for the whole household and children. This will be measured in g/day*child. The investigators will ask #times/week eachstaple was consumed as well as the average portion size consumed each time (g).The caregiver will provide information about the child's frequency of consumption over the past week for each food group.
Assessment of the nutritional adequacy of Nigerien children | 3 years
  Nutritional status of children in the household will be assessed using theFood Consumption Score Nutritional Quality Analysis (FCS-N) which wasbased on country-specific food groups. Food groups are orange fruits,orange vegetables, other fruits, eggs, dairy, organ meats, meat, fish,grains and legumes. Example of food items in the FCS-N assessment will be corroborated by a Nigerien maternal and child health expert. This will be measured in #times/week each food group was consumed.
Nutritional impact of a fortified cereal-based product for the improvement of micronutrient deficiencies among children aged 24-60 months. | 3 months
  Fortified flour consumption will be assessed by fortified flours intake(g/child*day). Micronutrient contribution will calculated by multiplying the amount of flour consumed/child * (mg zinc/g flour), (mg iron/g flour) and(ug RAE vitamin A/g flour).

CONTACTS AND LOCATIONS:
Overall Officials: Bruce R Hamaker, PhD, Principal Investigator — Purdue University
Locations (1):
- INRAN, Niamey, Niger

IPD SHARING:
Plan to Share IPD: No
No personal information was collected. There is not a plan to share data collected.